CLINICAL TRIAL: NCT02026531
Title: Novel MRI Techniques in the Evaluation of Pulmonary Vascular Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STH14070
Record Dates: First submitted 2012-06-08; First posted 2014-01-03 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3-Helium inhalation gas (Experimental): This is a pilot study. The aim is to recruit 20 patients who will all receive the product under investigation.
  Interventions: Other: 3-Helium gas

INTERVENTIONS:
Other: 3-Helium gas — 3-Helium gas for MRI contrast

SUMMARY:
The diagnosis of a patient with pulmonary hypertension (PH) requires many investigations. At present cardiac catheterisation is the cornerstone investigation in these patients where it is used to establish disease severity and estimate prognosis. It is an invasive procedure which is expensive and not without risk to the patient. Despite the multitude of tests performed, identifying those patients with PH who have a poor diagnosis can be difficult. The aim of this study is to improve the assessment of patients with PH using novel magnetic resonance techniques.

ELIGIBILITY:
Inclusion Criteria:

* All cases referred to the clinic for assessment for possible pulmonary hypertension.

Exclusion Criteria:

* patients with a cardiac pacemaker or retained temporary pacing wire
* patients with aneurysm clip
* non MRI compatible heart valve prosthesis
* intra orbital metalic foreign body
* pregnancy
* metal prosthesis/spinal rods
* retained shrapnel
* cochlear implants/bladder stimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
pulmonary artery diameter (mm) | up to 3 months
  Three-dimensional MRI imaging will be used to acquire cardiac dimensions and anatomical ventilation distribution as well as regional partial pressures of oxygen in the lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Elliot, MBChB MRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Pulmonary Vascular Disease Unit, Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom